CLINICAL TRIAL: NCT06438055
Title: Clinical Treatment of Refractory Breast Cancer Based on Organoid Drug Sensitivity Results
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Kingbio Medical (Beijing) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJBCPDO01
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Refractory Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Organoid-Guided therapy (Experimental): All patients will be included in a single-arm. Participants will undergo biopsy of tumor tissue for subsequent organoid generation and drug sensitivity tests.
  Interventions: Other: Chemotherapy and targeted-therapy guided by organoid drug sensitivity test

INTERVENTIONS:
Other: Chemotherapy and targeted-therapy guided by organoid drug sensitivity test — This study conducts drug sensitivity tests on various clinically approved drugs. The most sensitive drug for the patient is selected for treatment. This study aims to evaluate the clinical effectiveness of treatment plans guided by organoid drug sensitivity tests.

SUMMARY:
This study aims to enroll refractory breast cancer patients. Patient-derived organoid will be established, and drug sensitivity test will be conducted to intervene in the selection of clinical treatment plans. Efficacy evaluation and prognosis analysis will also be conducted. It is hoped that this study will provide a basis for the development of personalized treatment plans.

DETAILED DESCRIPTION:
Forty patients with refractory breast cancer who met the inclusion criteria were enrolled in the study after signing an informed consent form. Tumor samples were obtained through clinical puncture, and qualified samples were subjected to organoid modeling. Perform drug sensitivity test on the established breast cancer organoids. The drugs used are all that have been marketed and applied in clinical practice. According to the results of organoid drug sensitivity analysis, the patient received a treatment plan with relatively sensitive drugs. Follow up prognostic data and relevant clinical information of enrolled patients, conduct statistical analysis on the consistency between drug sensitivity test results and patient treatment response, and evaluate the clinical effectiveness of treatment plans guided by organoid drug sensitivity results.

ELIGIBILITY:
Inclusion Criteria:

1. Female, aged ≥ 18 years and ≤ 75 years old;
2. Breast cancer confirmed by histology or cytology;
3. One of the following two conditions shall be met: a) Operable breast cancer: Recurrent progression during adjuvant therapy; or the time from initial treatment to the onset of disease progression is less than or equal to 2 years; b) Non-operable breast cancer: patients who have changed two line treatment plans within 6 months;
4. Being able to obtain sufficient fresh tissue specimens for organoid establishment through puncture;
5. Expected survival time ≥ 3 months;
6. The patient voluntarily joined this study and signed an informed consent form (ICF), with good compliance and cooperation in follow-up.

Exclusion Criteria:

1. Pregnant and lactating women;
2. Patients who have clinically significant (i.e. active) heart disease (such as congestive heart failure, symptomatic coronary artery disease, arrhythmia, etc.) or myocardial infarction within the past 12 months;
3. Individuals with a history of abuse of psychotropic drugs who are unable to quit or have mental disorders;
4. The researchers believe that patients are not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 1-2 years
  Percentage of patient's measurable disease who have achieved either complete response (CR) or partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Progressive free survival | 1-2 years
  The time from initiation of treatment to the occurrence of disease progression or death.
Overall survival time | 2 years
  The time from the date of randomization to the date of death for any cause. Patients will be followed until their date of death or until final database closure.

CONTACTS AND LOCATIONS:
Overall Officials: Yehui Shi, PhD, Principal Investigator — Tianjin Cancer Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cao W, Chen HD, Yu YW, Li N, Chen WQ. Changing profiles of cancer burden worldwide and in China: a secondary analysis of the global cancer statistics 2020. Chin Med J (Engl). 2021 Mar 17;134(7):783-791. doi: 10.1097/CM9.0000000000001474. PMID 33734139
- [Background] Lei S, Zheng R, Zhang S, Chen R, Wang S, Sun K, Zeng H, Wei W, He J. Breast cancer incidence and mortality in women in China: temporal trends and projections to 2030. Cancer Biol Med. 2021 May 18;18(3):900-9. doi: 10.20892/j.issn.2095-3941.2020.0523. PMID 34002584
- [Background] Potter DA, Herrera-Ponzanelli CA, Hinojosa D, Castillo R, Hernandez-Cruz I, Arrieta VA, Franklin MJ, Yee D. Recent advances in neoadjuvant therapy for breast cancer. Fac Rev. 2021 Jan 4;10:2. doi: 10.12703/r/10-2. eCollection 2021. PMID 33659921
- [Background] Loibl S, Poortmans P, Morrow M, Denkert C, Curigliano G. Breast cancer. Lancet. 2021 May 8;397(10286):1750-1769. doi: 10.1016/S0140-6736(20)32381-3. Epub 2021 Apr 1. PMID 33812473
- [Background] Gralow JR, Burstein HJ, Wood W, Hortobagyi GN, Gianni L, von Minckwitz G, Buzdar AU, Smith IE, Symmans WF, Singh B, Winer EP. Preoperative therapy in invasive breast cancer: pathologic assessment and systemic therapy issues in operable disease. J Clin Oncol. 2008 Feb 10;26(5):814-9. doi: 10.1200/JCO.2007.15.3510. PMID 18258991
- [Background] Seidlitz T, Merker SR, Rothe A, Zakrzewski F, von Neubeck C, Grutzmann K, Sommer U, Schweitzer C, Scholch S, Uhlemann H, Gaebler AM, Werner K, Krause M, Baretton GB, Welsch T, Koo BK, Aust DE, Klink B, Weitz J, Stange DE. Human gastric cancer modelling using organoids. Gut. 2019 Feb;68(2):207-217. doi: 10.1136/gutjnl-2017-314549. Epub 2018 Apr 27. PMID 29703791
- [Background] Eiraku M, Watanabe K, Matsuo-Takasaki M, Kawada M, Yonemura S, Matsumura M, Wataya T, Nishiyama A, Muguruma K, Sasai Y. Self-organized formation of polarized cortical tissues from ESCs and its active manipulation by extrinsic signals. Cell Stem Cell. 2008 Nov 6;3(5):519-32. doi: 10.1016/j.stem.2008.09.002. PMID 18983967
- [Background] Romero-Calvo I, Weber CR, Ray M, Brown M, Kirby K, Nandi RK, Long TM, Sparrow SM, Ugolkov A, Qiang W, Zhang Y, Brunetti T, Kindler H, Segal JP, Rzhetsky A, Mazar AP, Buschmann MM, Weichselbaum R, Roggin K, White KP. Human Organoids Share Structural and Genetic Features with Primary Pancreatic Adenocarcinoma Tumors. Mol Cancer Res. 2019 Jan;17(1):70-83. doi: 10.1158/1541-7786.MCR-18-0531. Epub 2018 Aug 31. PMID 30171177
- [Background] Li M, Izpisua Belmonte JC. Organoids - Preclinical Models of Human Disease. N Engl J Med. 2019 Feb 7;380(6):569-579. doi: 10.1056/NEJMra1806175. No abstract available. PMID 30726695
- [Background] Sachs N, de Ligt J, Kopper O, Gogola E, Bounova G, Weeber F, Balgobind AV, Wind K, Gracanin A, Begthel H, Korving J, van Boxtel R, Duarte AA, Lelieveld D, van Hoeck A, Ernst RF, Blokzijl F, Nijman IJ, Hoogstraat M, van de Ven M, Egan DA, Zinzalla V, Moll J, Boj SF, Voest EE, Wessels L, van Diest PJ, Rottenberg S, Vries RGJ, Cuppen E, Clevers H. A Living Biobank of Breast Cancer Organoids Captures Disease Heterogeneity. Cell. 2018 Jan 11;172(1-2):373-386.e10. doi: 10.1016/j.cell.2017.11.010. Epub 2017 Dec 7. PMID 29224780
- [Background] Dekkers JF, Whittle JR, Vaillant F, Chen HR, Dawson C, Liu K, Geurts MH, Herold MJ, Clevers H, Lindeman GJ, Visvader JE. Modeling Breast Cancer Using CRISPR-Cas9-Mediated Engineering of Human Breast Organoids. J Natl Cancer Inst. 2020 May 1;112(5):540-544. doi: 10.1093/jnci/djz196. PMID 31589320
- [Background] Chen P, Zhang X, Ding R, Yang L, Lyu X, Zeng J, Lei JH, Wang L, Bi J, Shao N, Shu D, Wu B, Wu J, Yang Z, Wang H, Wang B, Xiong K, Lu Y, Fu S, Choi TK, Lon NW, Zhang A, Tang D, Quan Y, Meng Y, Miao K, Sun H, Zhao M, Bao J, Zhang L, Xu X, Shi Y, Lin Y, Deng C. Patient-Derived Organoids Can Guide Personalized-Therapies for Patients with Advanced Breast Cancer. Adv Sci (Weinh). 2021 Nov;8(22):e2101176. doi: 10.1002/advs.202101176. Epub 2021 Oct 4. PMID 34605222
- [Background] Chica-Parrado MR, Godoy-Ortiz A, Jimenez B, Ribelles N, Barragan I, Alba E. Resistance to Neoadjuvant Treatment in Breast Cancer: Clinicopathological and Molecular Predictors. Cancers (Basel). 2020 Jul 22;12(8):2012. doi: 10.3390/cancers12082012. PMID 32708049
- [Background] Drost J, Clevers H. Organoids in cancer research. Nat Rev Cancer. 2018 Jul;18(7):407-418. doi: 10.1038/s41568-018-0007-6. PMID 29692415
- [Background] Norman M, Rivers C, Lee YB, Idris J, Uney J. The increasing diversity of functions attributed to the SAFB family of RNA-/DNA-binding proteins. Biochem J. 2016 Dec 1;473(23):4271-4288. doi: 10.1042/BCJ20160649. PMID 27888239
- [Background] Hashimoto T, Matsuda K, Kawata M. Scaffold attachment factor B (SAFB)1 and SAFB2 cooperatively inhibit the intranuclear mobility and function of ERalpha. J Cell Biochem. 2012 Sep;113(9):3039-50. doi: 10.1002/jcb.24182. PMID 22566185
- [Background] Hutter K, Lohmuller M, Jukic A, Eichin F, Avci S, Labi V, Szabo TG, Hoser SM, Huttenhofer A, Villunger A, Herzog S. SAFB2 Enables the Processing of Suboptimal Stem-Loop Structures in Clustered Primary miRNA Transcripts. Mol Cell. 2020 Jun 4;78(5):876-889.e6. doi: 10.1016/j.molcel.2020.05.011. PMID 32502422
- [Background] Hammerich-Hille S, Bardout VJ, Hilsenbeck SG, Osborne CK, Oesterreich S. Low SAFB levels are associated with worse outcome in breast cancer patients. Breast Cancer Res Treat. 2010 Jun;121(2):503-9. doi: 10.1007/s10549-008-0297-6. Epub 2009 Jan 10. PMID 19137425
- [Background] Zhen H, Yao Y, Yang H. SAFB2 Inhibits the Progression of Breast Cancer by Suppressing the Wnt/beta-Catenin Signaling Pathway via NFAT5. Mol Biotechnol. 2023 Sep;65(9):1465-1475. doi: 10.1007/s12033-022-00649-z. Epub 2023 Jan 18. PMID 36652182